CLINICAL TRIAL: NCT00246259
Title: An Open-Label Randomized Trial Comparing Risperdal Consta With Oral Antipsychotic Care in the Treatment of Early Psychosis
Brief Title: A Trial Comparing Risperidone Long-Acting Injection With Oral Antipsychotic in the Treatment of Early Psychosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005959; RISSCH4056
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Results first posted 2013-11-12 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Psychotic Disorders
Keywords: Schizophrenia; Schizoaffective disorder; Schizophreniform disorder; Risperidone; Risperdal Consta
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Antipsychotic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risperidone long-acting injection (LAI) (Experimental): Risperidone LAI 25 mg, 37.5 mg or 50 mg intramuscular injection will be administered every 2 weeks as per Investigator's discretion. An oral atypical antipsychotic will also be administered in the first 3 weeks following initiation of Risperidone LAI, and for a maximum of 3 weeks following a dose increase.
  Interventions: Drug: Risperidone long-acting injection (LAI)
- Oral Antipsychotic (Active Comparator): Oral antipsychotic (new or current treatment) will be administered in which daily dose range permitted will be risperidone 6 mg; olanzapine 20 mg; quetiapine 800 mg. Participants will be switched to another oral therapy as per Investigator's discretion.
  Interventions: Drug: Oral Antipsychotic

INTERVENTIONS:
Drug: Risperidone long-acting injection (LAI) — Risperidone LAI 25 mg, 37.5 mg or 50 mg intramuscular injection will be administered every 2 weeks as per Investigator's discretion.
  Arms: Risperidone long-acting injection (LAI)
Drug: Oral Antipsychotic — Oral antipsychotic (new or current treatment) will be administered in which daily dose range permitted will be risperidone 6 mg; olanzapine 20 mg; quetiapine 800 mg.
  Arms: Oral Antipsychotic

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety and tolerability of risperidone long-acting injection (LAI) versus oral antipsychotics in participants with recent onset psychosis (abnormal thinking and/or hallucinations).

DETAILED DESCRIPTION:
This is an open-label (all people know identity of intervention), randomized (the study drug is assigned by chance), multicenter (conducted in more than 1 center), and exploratory study in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality) or schizoaffective disorder (mixed psychiatric disorder relating to complex psychotic state that has features of both schizophrenia and mood disorder). Duration of this study will be 24 months. Study assessment visits will be conducted at Screening, Baseline, Week 2, every 4 weeks till Week 22, at Week 28, every 12 weeks till Week 88 and at Week 104. All eligible participants will receive either risperidone long acting injection 25 milligram (mg) intramuscularly (into the muscle) along with their current oral medication (atypical antipsychotic - risperidone, quetiapine, olanzapine) or only their current oral medication. Efficacy will be evaluated primarily by Positive and Negative Syndromes Scale (PANSS), time to relapse and Social and Occupational Functioning Assessment Scale (SOFAS). Participants's safety will be evaluated throughout the study mainly by Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Rating Scale (BARS), and Simpson Angus Scale (SAS).

ELIGIBILITY:
Inclusion Criteria:

* In-patients or out-patients
* Primary Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) diagnosis of schizophrenia, schizophreniform disorder or schizoaffective disorder for no longer than 3 years after diagnosis and treatment of a psychotic illness
* Positive and Negative Syndrome Scale (PANSS) score of 60-120 at Visit 1 and 2
* Currently on monotherapy atypical antipsychotic treatment below local label guidelines or treatment naive
* Able to complete self-assessments in either English or French

Exclusion Criteria:

* Current primary Axis-1 diagnosis other than schizophrenia, schizophreniform disorder or schizoaffective disorder, according to DSM-IV
* Current drug or alcohol dependence
* Treatment with a depot antipsychotic within 3 months of study start
* Confirmed or suspected history of lack of tolerability, hypersensitivity or allergy to risperidone
* Risperidone non-responders (based on evidence of adequate trial of treatment)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2004-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (11):
- Canada (11):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Dartmouth, Nova Scotia
  - Greater Sudbury, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Markham, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Verdun, Quebec

REFERENCES:
- See also: An Open-label Randomized Trial Comparing RISPERDAL*CONSTA* With Oral Antipsychotic Care in the Treatment of Early Psychosis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=366&filename=CR005959_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone Long-acting Injection (LAI): Risperidone LAI 25 mg, 37.5 mg or 50 mg intramuscular injection was administered every 2 weeks as per Investigator's discretion. An oral atypical antipsychotic was administered in the first 3 weeks following initiation of Risperidone LAI, and for a maximum of 3 weeks following a dose increase.
- Oral Antipsychotic: Oral antipsychotic (new or current treatment) was administered in which daily dose range permitted was risperidone 6 mg; olanzapine 20 mg; quetiapine 800 mg. Participants switched to another oral therapy as per Investigator's discretion.
Period: Overall Study
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Started | 44 | 41
Eligible for Intent-to-treat (ITT) | 42 | 35
Completed | 16 | 15
Not Completed | 28 | 26
Not completed — Other | 3 | 3
Not completed — Not stable by Week 18 | 2 | 1
Not completed — Participant non-compliant | 4 | 9
Not completed — Lack of Efficacy | 2 | 2
Not completed — Investigator withdrew participant | 2 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 5 | 1
Not completed — randomly assigned, not eligible for ITT | 2 | 6

BASELINE CHARACTERISTICS:
Population: Analysis was based on the Intent-to-treat (ITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic | Total
Number analyzed (Participants) | 42 | 35 | 77
Age Continuous [Mean (Standard Deviation); unit: Years] | 22.5 (3.12) | 23.0 (2.93) | 22.7 (3.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 104 or Last Reported Visit (LRV)
Description: The PANSS provides a total score (sum of the scores of all 30 items) and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Baseline, Week 104 or LRV
Population: Intent-to-treat (ITT) analysis population included all the participants who received at least 3 doses of risperidone or 6 weeks of their oral antipsychotic, and had at least 1 post-baseline efficacy assessment. One participant was missing as reported in oral antipsychotic arm. 'n' = participants evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 42 | 35
Units on a scale
  Baseline (n=42, 35) | 80.6 (12.22) | 79.7 (12.47)
  Change at Week 104 or LRV (n=42, 34) | -18.1 (22.48) | -17.7 (16.45)

2. Primary Outcome: Time to Relapse
Description: Time to relapse was calculated from the start of the maintenance phase to date of relapse according to Csernansky: "Psychiatric hospitalization; increased level of psychiatric care from start of maintenance period and 25 percent increase in total PANSS score from first maintenance visit, or 10 points increase where PANSS at start of maintenance period was 40 or less; deliberate self-injury, suicidal or homicidal ideation; violent to others; property damage; or substantial clinical deterioration, defined as Clinical Global Impression of Change (CGI-C) score of 6 (much worse)".
Time Frame: Week 10 (post-stability) up to Week 104 or LRV
Population: The ITT analysis population included all the participants who received at least 3 doses of risperidone or 6 weeks of their oral antipsychotic, and had at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 42 | 35
Weeks | 80.5 (6.3) | 79.5 (4.1)

3. Primary Outcome: Change From Baseline in Social and Occupational Functioning Assessment Scale (SOFAS) at Week 104 or LRV
Description: The SOFAS focused exclusively on participants' level of social and occupational functioning. The SOFAS is a 100 point single item scale that rates functioning of a participant. The scale values range from 1=most impaired to 100=healthiest individual. The scale also includes a rating point of 0=missing information.
Time Frame: Baseline, Week 104 or LRV
Population: The ITT analysis population included all the participants who received at least 3 doses of risperidone or 6 weeks of their oral antipsychotic, and had at least 1 post-baseline efficacy assessment. Here 'n' = participants evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 42 | 35
Units on a scale
  Baseline (n=42, 35) | 53.4 (11.23) | 49.5 (12.93)
  Change at Week 104 or LRV (n=34, 28) | 4.6 (16.82) | 9.5 (15.24)

4. Secondary Outcome: Change From Baseline in Calgary Depression Symptom Scale (CDSS) Score at Week 104 or LRV
Description: Co-morbid depressive symptoms are evaluated by change in CDSS Score which was developed to assess symptoms of depression in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self). It consists of 9 items, each scored from 0 (absent) to 3 (severe). The total score is a sum of the scores of each item and may range from 0 to 27. Higher score more severe pathology. Data presented here represents the change from baseline to endpoint.
Time Frame: Baseline, Week 104 or LRV
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 42 | 35
Units on a scale
  Baseline (n=42, 35) | 3.7 (3.44) | 3.5 (2.80)
  Change at Week 104 or LRV (n=34, 28) | 0.1 (5.38) | -1.0 (3.12)

5. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) at Week 104 or LRV
Description: Co-morbid symptoms of mania are evaluated by change in YMRS Score which is an 11-item scale to assess symptoms of mania, Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 (the least) to 60 (the worst).
Time Frame: Baseline, Week 104 or LRV
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 42 | 35
Units on a scale
  Baseline (n=42,35) | 4.0 (4.02) | 4.3 (4.03)
  Change at Week 104 or LRV (n=34,28) | -1.1 (4.35) | -1.5 (3.33)

6. Secondary Outcome: Change From Baseline Hamilton Anxiety Scale (HAM-A) Total Score at Week 104 or LRV
Description: The HAM-A is a 14-item scale designed to measure anxiety in individuals. Each question reflects a symptom of anxiety and physical as well as mental symptoms are represented. The answers range from 0 which signifies a complete lack of that symptom to 4, which indicates a very severe show of anxiety with that symptom. Total score ranges from 0 to 56. Lower score indicates less affected.
Time Frame: Baseline, Week 104 or LRV
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 42 | 35
Units on a scale
  Baseline (n=42, 35) | 7.2 (5.94) | 7.3 (4.66)
  Change at Week 104 or LRV (n=34, 28) | -0.8 (6.23) | -2.9 (4.98)

7. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined according to Csernansky: "Psychiatric hospitalization; increased level of psychiatric care from start of maintenance period and 25 percent increase in total PANSS score from first maintenance visit, or 10 points increase where PANSS at start of maintenance period was 40 or less; deliberate self-injury, suicidal or homicidal ideation; violent to others; property damage; or substantial clinical deterioration, defined as CGI-C score of 6 (much worse)".
Time Frame: Week 10 (post-stability) up to Week 104 or LRV
Population: The ITT analysis population included all the participants who received at least 3 doses of risperidone or 6 weeks of their oral antipsychotic, and had at least 1 post-baseline efficacy assessment. Here 'N' (number of participants analyzed) = participants evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 32 | 31
Percentage of participants | 34.4 | 16.1

8. Secondary Outcome: Number of Participants With Cognitive Assessment Using Trail A
Description: Cognitive assessments were done using Trail test A which measured variety of functions, including motor speed, visual scanning, attention and visual motor integration. Participants must connect numbered circles in a variety of orders.
Time Frame: Week -2, 104 or LRV
Population: The ITT population included all participants who received at least 3 doses of risperidone or 6 weeks of oral antipsychotic, and had at least 1 post-baseline efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 42 | 35
Participants
  Week -2 (0-26 seconds) | 13 | 14
  Week -2 (27-39 seconds) | 16 | 9
  Week -2 (40-51 seconds) | 6 | 4
  Week -2 (52+ seconds) | 6 | 6
  Week -2 (Not reported) | 1 | 2
  Week 104 (0-26 seconds) | 15 | 16
  Week 104 (27-39 seconds) | 9 | 7
  Week 104 (40-51 seconds) | 4 | 3
  Week 104 (52+ seconds) | 2 | 2
  Week 104 (Not reported) | 12 | 7

9. Secondary Outcome: Number of Participants With Cognitive Assessments Using Trail B
Description: Cognitive assessments were done using Trail test B, which measured variety of functions, including motor speed, visual scanning, attention and visual motor integration. In Trail B, 2 sets of circles contain numbers and letters, and the participant must connect them in alternating order. Trail B is also a measure of executive functions as it requires planning and decision-making.
Time Frame: Week -2, 104 or LRV
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 42 | 35
Participants
  Week -2 (0-65 Seconds) | 17 | 12
  Week -2 (66-85 seconds) | 8 | 5
  Week -2 (86-120 seconds) | 8 | 3
  Week -2 (121+ seconds) | 8 | 13
  Week -2 (Not reported) | 1 | 2
  Week 104 (0-65 seconds) | 17 | 16
  Week 104 (66-85 seconds) | 7 | 4
  Week 104 (86-120 seconds) | 4 | 5
  Week 104 (121+ seconds) | 2 | 3
  Week 104 (Not reported) | 12 | 7

10. Secondary Outcome: Total Words Score Over Time
Description: Controlled Word Association Test (COWAT) was used to assess verbal fluency. Participants are given 3 different letters of the alphabet and asked to say as many words beginning with each letter within a controlled time. Participants are then asked to identify as many words as possible in 3 different categories (animals, fruits and vegetables) within a specified period of time. The total score is a sum of all three categories scores. The total score ranges from 0-90, the higher the score the higher the verbal fluency.
Time Frame: Baseline, Week 104 or LRV
Population: The ITT population:all participants who received at least 3 doses of risperidone or 6 weeks of oral antipsychotic, and had at least 1 post-baseline efficacy assessment. Here 'N' signifies participants evaluable for this measure and 'n' signifies participants evaluable at each time point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 40 | 31
Units on a scale
  Baseline (n=40, 31) | 62.4 (19.06) | 59.9 (16.49)
  Week 104 or LRV (n=30, 28) | 63.1 (17.81) | 65.4 (18.50)

11. Secondary Outcome: Change From Baseline in Drug Attitude Inventory (DAI-10) Score at Week 104 or LRV
Description: The DAI, a 10-item scale to assess how the attitude of schizophrenia participants toward their medications may affect compliance. Respondents indicate 'true' or 'false' for each item. An overall calculated score ranged from -10 to 10, where a positive score indicated a positive subjective response (compliant), a negative score indicated non-compliance. Change: score at observation minus score at baseline.
Time Frame: Up to Week 104 or LRV
Population: The ITT analysis population included all the participants who received at least 3 doses of risperidone or 6 weeks of their oral antipsychotic, and had at least 1 post-baseline efficacy assessment. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 33 | 27
Units on a scale | -0.1 (2.08) | -0.2 (2.71)

12. Secondary Outcome: Change From Baseline in Standardized Mental Component Scale Score in Short Form 36 (SF-36) at Week 104 or LRV
Description: The SF-36 is a survey of participant health. It calculates two standardized scales: the standardized mental component scale and the standardized physical component scale. The standardized scales are calculated as weighted sums of the 8 scores, which are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Each item is scored on a 0-100 range; and standardized mental component scale score is calculated as weighted average of individual item scores on a 0-100 range, where 100 signify highest level of functioning. The change from baseline in mental component scale score was reported.
Time Frame: Up to Week 104 or LRV
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 34 | 29
Units on a scale | 0.6 (14.95) | 4.7 (12.66)

13. Other Pre Specified Outcome: Barnes Akathisia Rating Scale (BARS) Global Clinical Assessment
Description: The BARS evaluates akathisia (feeling of restlessness) associated with the use of antipsychotic medications, including an objective and a subjective component plus a global impression. Components are rated on a scale of 0 (normal or absence of restlessness)-3 (intense restlessness) and 0 (absent)-5 (severe akathisia) for the global clinical assessment. Number of participants in each global clinical assessment scale are reported.
Time Frame: Baseline, Week 104 or LRV
Population: Analysis population included all randomly assigned participants. Here 'n' signifies participants evaluable at each time point for each treatment arm, respectively.
Measure: Number; unit: Participants
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 42 | 35
Participants
  Baseline: Absent (n=42,35) | 29 | 21
  Baseline: Questionable (n=42,35) | 11 | 8
  Baseline: Mild Akathisia (n=42,35) | 2 | 6
  Baseline: Moderate Akathisia (n=42,35) | 0 | 0
  Baseline: Marked Akathisia (n=42,35) | 0 | 0
  Week 104: Absent (n=35,29) | 21 | 25
  Week 104: Questionable (n=35,29) | 7 | 2
  Week 104: Mild Akathisia (n=35,29) | 6 | 2
  Week 104: Moderate Akathisia (n=35,29) | 1 | 0
  Week 104: Marked Akathisia (n=35,29) | 0 | 0

14. Other Pre Specified Outcome: Simpson Angus Scale (SAS)
Description: The SAS is a 10-item scale used to measure the symptoms of parkinsonism (slow movements) or parkinsonian side-effects related to the use of antipsychotic medications. The 10 items are rated on a 5-point scale (0=complete absence, 4=extreme presence) after a brief neurological examination and observation of the participants' gait (slow, shuffling walk). Total score is sum of individual item scores (range 0 to 40); higher score indicates more affected.
Time Frame: Baseline, Week 104 or LRV
Population: Analysis population included all randomly assigned participants. Here 'N' (Number of Participants Analyzed) signifies participants who were evaluable for this measure and 'n' signifies participants evaluable at each time point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 42 | 34
Units on a scale
  Baseline (n=42,34) | 1.1 (1.90) | 1.2 (1.61)
  Week 104 (n=34,29) | 1.0 (1.77) | 1.0 (2.10)

15. Other Pre Specified Outcome: Abnormal Involuntary Movement Scale (AIMS)
Description: The AIMS is a 12-item scale to provide a numeric measure to the observed abnormal movements in different parts of the body. Information is collected after a brief neurological examination and is scored on a 5-point scale (0=none, 4=severe). Ten items are scored in a 5-point scale (0 = none/normal, 4 = severe) which evaluates abnormal movements in three main anatomic areas (orofacial area, extremities, and trunk). Two items are yes/no questions regarding dental status. Total scores range from 0 to 42 with higher values indicating more severity.
Time Frame: Baseline, Week 104 or LRV
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Number analyzed (Participants) | 42 | 35
Units on a scale
  Baseline (n=42,35) | 1.1 (2.07) | 0.8 (1.35)
  Week 104 (n=35,29) | 0.7 (1.66) | 0.7 (1.37)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 104
Arm/Group | Risperidone Long-acting Injection (LAI) | Oral Antipsychotic
Serious Adverse Events (participants affected / at risk) | 2/44 | 3/41
Other Adverse Events (participants affected / at risk) | 38/44 | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone Long-acting Injection (LAI) (N=44) | Oral Antipsychotic (N=41)
Alcoholism (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Skin laceration (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone Long-acting Injection (LAI) (N=44) | Oral Antipsychotic (N=41)
Palpitations (Cardiac disorders) | 2 | 1
Vision blurred (Eye disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 6 | 2
Stomach discomfort (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
Fatigue (General disorders) | 11 | 5
Bronchitis (Infections and infestations) | 2 | 3
Ear infection (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 2 | 2
Nasopharyngitis (Infections and infestations) | 9 | 7
Sinusitis (Infections and infestations) | 2 | 2
Hand fracture (Injury, poisoning and procedural complications) | 1 | 2
Blood cholesterol increased (Investigations) | 1 | 2
Blood prolactin increased (Investigations) | 5 | 0
Blood triglycerides increased (Investigations) | 2 | 3
Weight decreased (Investigations) | 0 | 2
Weight increased (Investigations) | 10 | 7
Increased appetite (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Akathisia (Nervous system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 8 | 5
Dyskinesia (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 15 | 5
Lethargy (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 3 | 3
Tremor (Nervous system disorders) | 3 | 1
Aggression (Psychiatric disorders) | 0 | 2
Agitation (Psychiatric disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 6 | 4
Depression (Psychiatric disorders) | 3 | 3
Depressive symptom (Psychiatric disorders) | 2 | 0
Hallucination (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 13 | 7
Psyshotic disorder (Psychiatric disorders) | 4 | 4
Restlessness (Psychiatric disorders) | 1 | 2
Amenorrhoea (Reproductive system and breast disorders) | 5 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 1
Galactorrhoea (Reproductive system and breast disorders) | 2 | 1
Gynaecomastia (Reproductive system and breast disorders) | 2 | 2
Sexual dysfunction (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less